CLINICAL TRIAL: NCT00051675
Title: An Open-Label, Multi-Dose, Phase I, Dose-Escalating Study of a Subcutaneously Administered Human-Engineered Monoclonal Antibody, ING-1(heMAb), in Subjects With Advanced Adenocarcinomas
Brief Title: Phase I Study of a Monoclonal Antibody for Treatment of Advanced Adenocarcinomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: XOMA (US) LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCA104
Record Dates: First submitted 2003-01-14; First posted 2003-01-16 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-09

CONDITIONS: Adenocarcinoma
Keywords: adenocarcinoma; monoclonal antibody
MeSH Terms: conditions — Adenocarcinoma

INTERVENTIONS:
Drug: ING-1(heMAb)

SUMMARY:
The purpose of this study is to evaluate the safety, immunogenicity, and tolerability of a monoclonal antibody administered subcutaneously in the treatment of advanced cancers of the ovary, breast, lung, prostate, colon or rectum that are either refractory to standard therapies or for which therapies that may potentially be of major benefit do not exist.

ELIGIBILITY:
Inclusion Criteria

1. Subject has adenocarcinomas of the ovary, breast, lung, prostate, colon or rectum.
2. Subject has an advanced metastatic adenocarcinoma that is either refractory to standard therapies or for which therapies that may potentially be of major benefit do not exist.
3. Subject has measurable lesions. Subjects with prostate cancer can have non-measurable lesions.
4. Subject may have prior radiation therapy if completed at least four weeks prior to study entry, the subject has recovered from the acute toxicities of that therapy, and measurable lesions are in a non-irradiated area.
5. Subject may have prior chemotherapy, cytokine therapy or immunotherapy if completed at least four weeks prior to study entry and the subject has recovered from the acute toxicities of that therapy.
6. Subjects with tumors responsive to hormone therapy may have prior hormonal therapy if completed at least four weeks prior to study entry. Hormonal therapy for prostate cancer may be continued but must not have been changed less than four weeks prior to study entry.
7. Subject has a performance status of 0 to 2 on the Eastern Cooperative Oncology Group (ECOG) scale.
8. Subject has an estimated life expectancy of at least 12 weeks.
9. Subject is at least 18 years of age.
10. Subject has adequate organ function defined as follows:

    * Hematologic:

      * Platelets 100 × 109/L
      * Hemoglobin 9.0 g/dL
      * Total WBC count 3.5 × 109/L
      * PT/INR and PTT are within institutional limits in subjects who are not receiving therapeutic anticoagulation or low dose anticoagulants to maintain venous catheter patency (subjects on anti-coagulant therapy are allowed).
    * Hepatic:

      * Bilirubin 2.0 mg/dL
      * Aspartate transaminase (AST) and alanine transaminase (ALT) 3 times the upper limit of normal (AST and ALT 5 times the upper limit of normal is acceptable if liver has tumor involvement and the elevation is due to tumor involvement)
    * Renal: Serum creatinine 1.5 mg/dL
    * Pancreatic: Amylase and lipase upper limit of the normal (ULN)
11. Signed informed consent form.
12. Male and female subjects with reproductive potential must use an approved contraceptive method.
13. Female subjects with reproductive potential must have a negative serum pregnancy test within seven days of study enrollment.

Exclusion Criteria

1. Subject has serious concomitant systemic disorders incompatible with the study.
2. Subject has used any other investigational agent within 30 days of study entry.
3. Subject is pregnant or lactating.
4. Subject has undergone a bone marrow transplant.
5. Subject is known to be HIV+ or to have any other recognized immunodeficiency disease. (Note: As the mechanism of action of ING-1(heMAb) is ADCC, subjects need to be immunocompetent).
6. Subject has a history of severe allergic or anaphylactic reactions to monoclonal antibodies or antibody fragments. (Note: For subjects who have received prior ING-1(heMAb), the HAHA titer should be negative.)
7. Subject has concurrent or prior malignancy, except for adequately-treated basal cell or squamous cell skin cancer, adequately-treated non-invasive carcinomas or other cancer from which the subject has been disease-free for at least two years.
8. Subject has an active auto-immune disease requiring chronic treatment.
9. Subject is using or has used immunosuppressive drugs such as cyclosporine, ACTH or corticosteroids within four weeks prior to enrollment.
10. Subject has brain metastases or a known history of brain metastases.
11. Subject has a history of alcoholism or chronic pancreatitis or a family history of acute or chronic pancreatitis.
12. Subject has hypertriglyceridemia ( Serum triglycerides 500 mg/dL).
13. Subject has a history of gall bladder disease or gallstones (post-cholecystectomy subjects are allowed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2002-07; Study Completion 2003-09

CONTACTS AND LOCATIONS:
Locations (1):
- Jack D. Weiler Hospital of the Albert Einstein College of Medicine, The Bronx, New York, United States